CLINICAL TRIAL: NCT03599778
Title: A Phase I/II Clinical Study to Compare Postoperative Chemotherapy of Oxaliplatin With Capecitabine（XELOX）Combined With APATINIB as Post-operative Chemotherapy in Locally Advanced Gastric Adenocarcinoma With D2 Dissection
Brief Title: XELOX Combined With Apatinib as Post-operative Chemotherapy in Locally Advanced Gastric Adenocarcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHTH-201
Record Dates: First submitted 2018-06-14; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Gastric Carcinoma
Keywords: apatinib; Gastric Carcinoma; post-operative chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): 8 cycles of postoperative XELOX regimen (capecitabine: 1000 mg/m2 bid d1-14 q3w, oxaliplatin: 130 mg/m2 d1 q3w) + apatinib'MTD(maximum tolerated dose)
  Interventions: Drug: Apatinib
- Control group (Active Comparator): 8 cycles of postoperative XELOX regimen (capecitabine: 1000 mg/m2 bid d1-14 q3w, oxaliplatin: 130 mg/m2 d1 q3w)
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — XELOX + apatinib's MTD
  Other Names: XELOX

SUMMARY:
To observe and evaluate the efficacy and safety of oxaliplatin with oapecitabine（XELOX）combined with apatinib as post-operative chemotherapy in locally advanced gastric adenocarcinoma with D2 dissection

DETAILED DESCRIPTION:
Stage 1 (phase I tolerance study) : 12 patients were enrolled in the dose-climbing study:According to the principle of dose-climbing test,todetermine the subjects' MTD, with the following three dose levels:

* Capecitabine: 1000 mg/m2 bid d1-14 q3w, oxaliplatin: 130 mg/m2 d1 q3w) + apatinib 250 mg, qd x180d; ②. Capecitabine: 1000 mg/m2 bid d1-14 q3w, oxaliplatin: 130 mg/m2 d1 q3w) + apatinib 375 mg, qd x180d; ③. Capecitabine: 1000 mg/m2 bid d1-14 q3w, oxaliplatin: 130 mg/m2 d1 q3w) + apatinib 500 mg, qd x180d;

Stage 2 (phase II exploratory study) :

①.Test group: subjects received 8 cycles of postoperative XELOX regimen (capecitabine: 1000 mg/m2 bid d1-14 q3w, oxaliplatin: 130 mg/m2 d1 q3w) + apatinib maximum tolerated dose

②.Control group: Subjects received 8 cycles of XELOX regimen after surgery (capecitabine: 1000 mg/m2 bid d1-14 q3w, oxaliplatin: 130 mg/m2 d1 q3w).

Eligible patients will receive 8 cycles of postoperative adjuvant therapy and will be followed up to death

ELIGIBILITY:
Inclusion Criteria:

1. ECOG score is 0-1;
2. Radical gastrectomy (D2, R0) for gastric cancer has been performed (more than 16 lymph nodes have been detected);
3. Postoperative histology confirmed gastric adenocarcinoma；
4. The pathological stage of gastric cancer is ⅢA-ⅢC stage (8th AJCC TNM);
5. Subjects' baseline blood routine and biochemical indicators meet the following standards:

   * ANC≥1.5×109/L;
   * Hb≥90g/L;
   * PLT≥100×109/L;
   * TBIL≤1.5×ULN;
   * ALT and AST≤2×ULN;
   * Cr≤1.5×ULN
   * INR：1.0～1.5; APTT is within the normal range
6. The electrocardiogram was basically normal before the first 4 weeks after admission, and there were no obvious clinical symptoms of heart disease;
7. Sign informed consent.

Exclusion Criteria:

1. Patients with severe hypertension and poor drug control;
2. Various factors that affect oral drugs such as (inability to swallow, complete or incomplete gastrointestinal obstruction, active gastrointestinal bleeding, perforation ) ;
3. Patients with previous bradycardia or prolonged QT interval;
4. Patients with postoperative gastrointestinal fistula and wound rupture;
5. Known allergy to capecitabine or oxaliplatin, or metabolic disorder;
6. Patients receiving preoperative chemotherapy, radiotherapy or targeted therapy before;
7. Patients Using other experimental drugs at the same time or joining in other clinical trials.
8. Patients with severe liver diseases (such as liver cirrhosis), nephropathy, respiratory diseases or chronic systemic diseases such as uncontrollable diabetes and hypertension; Clinical symptoms of heart disease,such as congestive heart failure,coronary heart disease symptoms, arrhythmia, hypertension,that hard to control,or having myocardial infarction attack in six months or cardiac insufficiency.
9. Patients with peripheral nervous system disorder or with a history of significant psychiatric disorder and central nervous system disorder;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3 months
  Disease-free survival (DFS) is defined as the time from the beginning of treatment to Disease recurrence or death due to Disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Xinyang He, master, Principal Investigator — Anhui Provincial Cancer Hospital
Locations (1):
- Anhui Provincial Cancer Hospital, Hefei, Anhui, China